CLINICAL TRIAL: NCT06020456
Title: Study of Genetic Factors Influencing the Factor VIII Response to Desmopressin in Carriers of Hemophilia A: the GIDEHAC Study
Brief Title: Genetic Factors of the Desmopressin Response in Carriers of Hemophilia A
Acronym: GIDEHAC
Status: Completed | Type: Observational
Sponsor: Groupe Maladies hémorragiques de Bretagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_GIDEHAC_01
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Carrier of Hemophilia A; Desmopressin; Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Variants Null: This group includes patients carrying a F8 variant with a major deleterious effect on the F8 gene (non-sense, intron 1 and 22 inversions, large deletions, small insertions/deletions leading to a frameshift and premature stop codon)
  Interventions: Drug: Desmopressin
- Variants No Null: This group includes patients carrying a F8 variant with a mild effect on the F8 gene (missense, splice modification, small nucleotide deletion in the intron 13, and variant in the promoter)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — For the 2 groups, all patients have received an intravenous DDAVP 0,3-0,4 µg/Kg infusion associated with pre/post-desmopressin measurements of plasma FVIII levels

SUMMARY:
Hemophilia A (HA) is a rare X-linked bleeding disorder caused by a deficiency in factor VIII (FVIII) affecting 1/5,000 males1. Carriers of HA are females carrying the pathogenic variant responsible for the familial HA at a heterozygous status. About 30% of HA carriers have low FVIII levels and can therefore have abnormal bleeding symptoms2,3. Such as males with moderate/mild HA, bleeding can be treated or prevented with either FVIII concentrates or desmopressin4,5. This drug acts as a vasopressin type 2-receptor (V2R) agonist that causes endothelial cells to rapidly secrete von Willebrand factor (VWF) and FVIII from Weibel-Palade bodies into the bloodstream6,7. However, the mechanism of action of post-DDAVP FVIII increase remains poorly understood in hemophilia A. One advantage of DDAVP is that it increases the level of endogenous FVIII, thus avoiding the need for potentially immunogenic exogenous FVIII. It is also cheaper than FVIII concentrates. Finally, it is more widely available in pharmacies in all hospitals with emergency rooms and surgical facilities.

The FVIII response profile to DDAVP in carriers appears quite similar to that seen in men with mild/moderate HA8-11. A post-DDAVP increase in the FVIII level of 2-4 fold the basal level is usually observed. This FVIII response presents an important inter-individual variation making it necessary to carry out a therapeutic test before its use for the anti-hemorrhagic treatment. The basal FVIII level logically conditions the intensity of the post-DDAVP FVIII peak. However, other factors influencing the post-DDAVP FVIII response are very likely. Unfortunately, few series describing the FVIII response to DDAVP in HA carriers have been reported to date and they included too small numbers of patients to precisely analyze the factors of variation in the post-DDAVP FVIII pharmacokinetics (PK). Candy et al did not find any difference depending on the severity of the pathogenic variants for HA or on the age11. However, this study was carried out in a cohort including only 17 patients, therefore too small for a reliable statistical analysis.

The GIDEHAC study (Genetic Influence of Desmopressin Efficacy in Hemophilia A Carriers) is a French study with the following objectives: the description of the post-DDAVP FVIII PK in a large retrospective cohort of HA carriers, the research of patients-related factors influencing this FVIII PK, and the building of predictive population- and Bayesian-based models.

DETAILED DESCRIPTION:
The GIDEHAC study is a French observational, retrospective, and multicentric study performed in carriers of hemophilia A of any age who have received the intravenous desmopressin in their French Hemophilia Treatment Centers (HTC).

Objectives of the GIDEHAC study:

* Description of the post-desmopressin (DDAVP) FVIII pharmacokinetics (PK) in a large retrospective cohort of patients with mild/moderate HA,
* Research of patients-related factors influencing this FVIII PK,
* Building of predictive population- and Bayesian-based models

Inclusion criteria:

* Females at any ages with a confirmed diagnosis of HA carriers based on the F8 gene analysis,
* Patients having received DDAVP during the last 10 years that was associated with dosages of FVIII before and just after DDAVP,
* Factor VIII levels measurements realized at least 2 times during the therapeutic test, just before the DDAVP infusion and 30 or 60 minutes after.

Exclusion criteria:

* Patients with an anti-factor VIII inhibitor,
* Refusal to participate in the study,
* Unable to understand the study's French letter of non-opposition and information.

Description of the DDAVP therapeutic tests:

The procedure of the DDAVP therapeutic test was identical for all investigator centers as recommended by international and French guidelines. DDAVP was so always administered intravenously at a dose of 0.3-0.4 μg.kg-1 diluted in 50 mL of saline solution over 30 minutes. The required hemostatic parameters are FVIII levels before and at least 30 or 60 minutes after the DDAVP infusion. Subsequent FVIII measurements performed at T2h, T4h and T6h after the infusion are also recorded during the test.

Collected data:

All data collected in this study were issued from the medical files at the moment of the DDAVP therapeutic test. They include:

* FVIII activity levels measured with a one-stage clotting assay from plasmas collected in 0.109 M sodium citrate (fresh or stored at -80°C). These FVIII levels were measured just before and after the DDAVP infusion (until 24 hours if available),
* The pathogenic variant of the F8 gene responsible for the familial HA,
* Blood group,
* DDAVP doses,
* Von Willebrand factor levels during the DDAVP test,
* Age,
* Weight,
* FVIII levels measured during pregnancies,
* The degree of familial link if relatives are included in this study.

Pharmacokinetic analyses The following FVIII and VWF pharmacokinetic parameters are calculated using a compartmental approach with non-linear models at mixed effect (MONOLIX software, v2021, Lixsoft): basal FVIII and post-DDAVP FVIII peak (highest level measured after DDAVP administration), FVIII recovery (recFVIII = peak FVIII / basal FVIII), FVIII half-life (FVIII T1/2), FVIII clearance, FVIII area under the curve (FVIII AUC), and duration with FVIII ≥0.5 and 0.8 IU.dL-1.

Scores measuring the FVIII response to DDAVP

For qualitative assessment of the biological response to DDAVP, criteria previously reported by Stoof et al were used:

* The absolute response was either "complete" (peak FVIII ≥0.5 IU.mL-1), "partial" (FVIII ≥0.3 - <0.5 IU.mL-1) or "null" (FVIII <0.3 IU.mL-1).
* The relative response was defined as "complete" (recFVIII >3), "partial" (recFVIII ≥2 - <3) or "null" (recFVIII <2).

ELIGIBILITY:
Inclusion Criteria:

* Females at any ages with a formal diagnosis of HA carriers based on the F8 genetics,
* Patients having received DDAVP during the last 10 years that was associated with dosages of FVIII before and just after DDAVP,
* Factor VIII levels measurements realized at least 2 times during the therapeutic test, just before the DDAVP infusion and 30 or 60 minutes after.

Exclusion Criteria:

* Patients with an anti-factor VIII inhibitor,
* Refusal to participate in the study,
* Unable to understand the study's French letter of non-opposition and information

Ages: 2 Years to 80 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The eligibility is based on the caryotype XX
Study Population: The study includes carriers of hemophilia A of any age who had a desmopressin therapeutic test during the last 10 years, associated with FVIII levels measurements before/after desmopressin.
  All procedures of the desmopressin therapeutic tests comprised an intravenous infusion of 0.3-0.4 μg.kg-1 diluted in 50 mL of saline solution over 30 minutes, associated with FVIII levels measured before and at least 30 or 60 minutes after the desmopressin infusion. Subsequent measurements performed at T2h, T4h and T6h after the infusion are also recorded during the test.
  All the data collected in this study were issued from the medical files including: pre/post desmopressin FVIII and VWF levels, F8 mutation, severity of the familial hemophilia A blood group, desmopressin doses, age, and weight.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the post-DDAVP FVIII peak in patients of the group "Null variants" vs "No Null variants" | FVIII levels 30-60 minutes after the DDAVP infusion
  Factor VIII levels measured with a chronometric one stage-assay 30 or 60 minutes after the DDAVP infusion
Comparison of the post-DDAVP FVIII recovery in patients of the group "Null variants" vs "No Null variants" | FVIII levels before and 30-60 minutes after the DDAVP infusion
  Factor VIII levels measured with a chronometric one stage-assay before (basal FVIII) the DDAVP infusion and 30 or 60 minutes after (FVIII peak). The FVIII recovery = ratio FVIII peak / basal FVIII
Comparison of the post-DDAVP FVIII clearance in patients of the group "Null variants" vs "No Null variants" | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  Factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion
Comparison of the post-DDAVP FVIII area under the curve (AUC) in patients of the group "Null variants" vs "No Null variants" | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  Factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion
Comparison of the post-DDAVP duration with FVIII normalized above 0.5 IU.dL-1 in patients of the group "Null variants" vs "No Null variants" | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  Factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion
Comparison of the post-DDAVP duration with FVIII normalized above 0.8 IU.dL-1 in patients of the group "Null variants" vs "No Null variants" | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  Factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion

SECONDARY OUTCOMES:
Influence of the age on the post-DDAVP FVIII peak | FVIII levels 30-60 minutes after the DDAVP infusion
  factor VIII levels measured with a chronometric one stage-assay 30 or 60 minutes after the DDAVP infusion
Influence of the age on the post-DDAVP FVIII recovery | FVIII levels before and 30-60 minutes after the DDAVP infusion
  Factor VIII levels measured with a chronometric one stage-assay before (basal FVIII) the DDAVP infusion and 30 or 60 minutes after (FVIII peak). The FVIII recovery = ratio FVIII peak / basal FVIII
influence of the age on the post-DDAVP FVIII area under the curve (AUC) | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  Factor VIII levels measured with a chronometric one stage-assay before (basal FVIII) the DDAVP infusion and 30 or 60 minutes after (FVIII peak). The FVIII recovery = ratio FVIII peak / basal FVIII
influence of the age on the post-DDAVP duration with FVIII normalized above 0.5 IU.dL-1 | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion
influence of the age on the post-DDAVP duration with FVIII normalized above 0.8 IU.dL-1 | Factor VIII levels were measured until 24 hours after the desmopressin infusion
  factor VIII levels measured with a chronometric one stage-assay before and after DDAVP until 24h post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Guillet, MD PhD, Principal Investigator — University-hospital of Rennes and Inserm U1085 (IRSET), Faculty of Medicine, University Rennes 1
Locations (12):
- France (12):
  - University hospital of Bordeaux, Bordeaux
  - University hospital of Brest, Brest
  - Hospices civils de Lyon, Bron
  - University hospital of Dijon, Dijon
  - University hospital of Bicêtre, Le Kremlin-Bicêtre
  - University hospital of Lille, Lille
  - Assistance publique hôpitaux de Marseille, Marseille
  - University hospital of Montpellier, Montpellier
  - University hospital of Nancy, Nancy
  - University hospital of Nantes, Nantes
  - University hospital of Rennes, Rennes
  - University hospital of Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Background] Seaman CD, Xavier F, Ragni MV. Hemophilia A (Factor VIII Deficiency). Hematol Oncol Clin North Am. 2021 Dec;35(6):1117-1129. doi: 10.1016/j.hoc.2021.07.006. Epub 2021 Aug 10. PMID 34389199
- [Background] Plug I, Mauser-Bunschoten EP, Brocker-Vriends AH, van Amstel HK, van der Bom JG, van Diemen-Homan JE, Willemse J, Rosendaal FR. Bleeding in carriers of hemophilia. Blood. 2006 Jul 1;108(1):52-6. doi: 10.1182/blood-2005-09-3879. Epub 2006 Mar 21. PMID 16551972
- [Background] Mannucci PM, Vicente V, Alberca I, Sacchi E, Longo G, Harris AS, Lindquist A. Intravenous and subcutaneous administration of desmopressin (DDAVP) to hemophiliacs: pharmacokinetics and factor VIII responses. Thromb Haemost. 1987 Dec 18;58(4):1037-9. PMID 3127916
- [Background] Leissinger C, Carcao M, Gill JC, Journeycake J, Singleton T, Valentino L. Desmopressin (DDAVP) in the management of patients with congenital bleeding disorders. Haemophilia. 2014 Mar;20(2):158-67. doi: 10.1111/hae.12254. Epub 2013 Aug 12. PMID 23937614
- [Background] van Galen KPM, d'Oiron R, James P, Abdul-Kadir R, Kouides PA, Kulkarni R, Mahlangu JN, Othman M, Peyvandi F, Rotellini D, Winikoff R, Sidonio RF. A new hemophilia carrier nomenclature to define hemophilia in women and girls: Communication from the SSC of the ISTH. J Thromb Haemost. 2021 Aug;19(8):1883-1887. doi: 10.1111/jth.15397. PMID 34327828
- [Background] Kaufmann JE, Vischer UM. Cellular mechanisms of the hemostatic effects of desmopressin (DDAVP). J Thromb Haemost. 2003 Apr;1(4):682-9. doi: 10.1046/j.1538-7836.2003.00190.x. PMID 12871401
- [Background] Kaufmann JE, Oksche A, Wollheim CB, Gunther G, Rosenthal W, Vischer UM. Vasopressin-induced von Willebrand factor secretion from endothelial cells involves V2 receptors and cAMP. J Clin Invest. 2000 Jul;106(1):107-16. doi: 10.1172/JCI9516. PMID 10880054
- [Background] Hews-Girard J, Rydz N, Lee A, Goodyear MD, Poon MC. Desmopressin in non-severe haemophilia A: Test-response and clinical outcomes in a single Canadian centre review. Haemophilia. 2018 Sep;24(5):720-725. doi: 10.1111/hae.13586. Epub 2018 Jul 13. PMID 30004154
- [Background] Kobrinsky NL, Watson CM, Cheang MS, Bishop AJ. Improved hemophilia A carrier detection by DDAVP stimulation of factor VIII. J Pediatr. 1984 May;104(5):718-24. doi: 10.1016/s0022-3476(84)80951-8. PMID 6425482
- [Background] Casonato A, Dannhauser D, Pontara E, Bertomoro A, Orazi B, Santarossa L, Zerbinati P, Girolami A. DDAVP infusion in haemophilia A carriers: different behaviour of plasma factor VIII and von Willebrand factor. Blood Coagul Fibrinolysis. 1996 Jul;7(5):549-53. PMID 8874865